CLINICAL TRIAL: NCT06854380
Title: Effect of Intralesional Injection of Corticosteroids Combined with Hyaluronidase in Treatment of Minimal Associated Pathological Lesions of Vocal Folds
Brief Title: Effect of Intralesional Injection of Corticosteroids Combined with Hyaluronidase in Treatment of Minimal Associated Pathological Lesions of Vocal Folds, Participants and Condition: Patients with Benign Vocal Fold Lesions, Intervention: Intralesional Injection Via Working Channel of Nasofiberscope
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD.24.12.933 - 29/12/2024
Record Dates: First submitted 2025-02-09; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Voice and Voice Disorders
MeSH Terms: conditions — Voice Disorders | interventions — Betamethasone; Hyaluronoglucosaminidase; Enzymes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group of patients suffering from dysphonia, laryngeal examination showed benign vocal fold lesions (Experimental)
  Interventions: Drug: Intralesional injection of steroids (betamethasone), (Betafos®) and hyaluronidase (enzyme), (Hynidase®) into benign vocal fold lesions by a naso-fiberscope with a side working channel(Storz 11001UD1)

INTERVENTIONS:
Drug: Intralesional injection of steroids (betamethasone), (Betafos®) and hyaluronidase (enzyme), (Hynidase®) into benign vocal fold lesions by a naso-fiberscope with a side working channel(Storz 11001UD1) — that this intervention is intralesional injection of glucocorticoid (betamethasone) and enzyme (hyaluronidase) via flexible fiberscope

SUMMARY:
Voice disorders encompass a wide range of pathologies that result in various degrees of voice impairment and decreased quality of life, Minimal Associated Pathological Lesions (MAPLs), include a group of non-malignant growths on the vocal folds like vocal fold nodules, polyps, papilloma, Reinke's oedema, polypoidal degeneration and cysts, The pathophysiology of MAPLs include abnormal inflammatory response to local trauma. Histologically, the superficial layer of the lamina propria shows oedema, fibrosis, fibrin and hemosiderin deposit, interstitial haemorrhage and inflammatory cell infiltration, Treatment options include voice therapy, intralesional steroid injections, and surgical. Although vocal function improves and lesion regresses by vocal hygiene advice and voice therapy, each patient receives two therapy sessions per week for about 3 months of voice treatment in the form of a holistic voice rehabilitation program. A total of 20 sessions are conducted, with each session lasting approximately 20 minutes; Which some patients find difficult.

Vocal folds (VFs) local steroid injection could bridge the therapeutic gap between conservative treatment and conventional micro laryngeal surgery (MLS), Steroids are thought to be useful for MAPLs as they share common histological features, including oedema, thick basement membrane, inflammation, and vessel wall thickness.

Steroids act by inhibiting both collagen deposition and collagen synthesis. Also, it acts by inhibiting fibroblastic proliferation and activity plus reduction of the extracellular matrix deposition.

Office-based vocal fold steroid injection (VFSI) can be performed through transoral, percutaneous and trans nasal routes, With several benefits Compared to MLS, it may be conducted in the office under local anaesthesia in about 20 minutes, saving high costs of general anaesthesia and hospital admission, decreasing lost workdays associated with recurrent voice therapy sessions.

Hyaluronidase (HAase) is a preparation of proteolytic enzyme. Its injection is indicated as an adjuvant in subcutaneous fluid administration for achieving hydration and for improving the dispersion and the absorption of injected drugs. HAase can be used in phono-surgery or in office applications. HAase has been useful in the following indications: (1) HA over-injection in the vocal fold after injection laryngoplasty, (2) treatment of Reinke's oedema and (3) in selected patients with acute vocal fold haemorrhage, improvement of the absorption of blood products. HAase appears to be useful in the office and the operative setting with minimal complications. There is a growing evidence in literature that using a steroid in combination with HAase maximizes the anti-inflammatory properties of the steroid and minimizes the side effects of steroid therapy.

Although voice therapy may be the first line of treatment for many benign vocal folds lesions, satisfactory outcomes are not obtained in some patients for many reasons. A patient would attend 20 to 25 sessions of voice therapy in order to show improvement and this would take 2 to 3 months.

Some patients, especially those from far residence, would find it difficult for them to comply to this relatively lengthy course of therapy, resulting in a number of drop out cases. Similarly, some professional voice users would hope to have their voice problem alleviated in a faster way. Moreover some patients show poor understanding of the procedure itself and hence could not implement it properly. For those reasons voice therapy may not be appropriate for those patients.

Based on previous background, we thought that intralesional injection of a combination of HAase and steroids into MAPls would not only provide a faster way for the patient to restore her/his normal voice but also would augment the effect of steroids by improving its delivery and dispersion into the lesion.

This is the first study to assess the effect of intralesional injection of a combination of steroid and HAase in treatment of MAPLs.

The aim of this study is to assess the effect of intralesional injection of minimal associated pathological lesions of the vocal folds by a combination of steroids and hyaluronidase in terms of subjective and objective voice outcomes and lesion regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with minimal associated pathological lesions and complaining of dysphonia and not fit for surgery.
* Patient not compliant to voice therapy (e.g. those from far residence).
* Patients who refuse voice therapy.
* Patient not responding to voice therapy.

Exclusion Criteria:

* Patients' refusal to be included in the study.
* Patients having any other laryngeal voice disorders.
* Patients not tolerating the naso-endoscopic examination.
* Patients having allergy to the injected material after doing intradermal allergy test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Auditory perceptual assessment of voice following a modified GRBAS scale (G: grade, R: roughness, B: breathiness, A: asthenia, S: strain), with 4 grades from 0 (normal) to 3 (severe dysphonia) for determining grade and character of dysphonia | 3 months from injection

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University - Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided